CLINICAL TRIAL: NCT03047785
Title: Is the Current Threshold for Diagnosis of "Abnormality", Including Non ST Elevation Myocardial Infarction, Using Raised Highly Sensitive Troponin Appropriate for a Hospital Population? The CHARIOT Study
Acronym: CHARIOT
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAR0516
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Highly sensitive troponin; Hospital population; 99th percentile; Upper limit of normal
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital population: All patients who have had a biochemistry blood tests requested at the trust will have a troponin blood level determined.

SUMMARY:
Currently when defining the upper limit of normal (ULN) or 99th percentile of a troponin assay manufacturer's use a healthy population traditionally aged 18-40. The 99th percentile value is the recommended value to use when diagnosing patients with an acute myocardial infarction. With the advent of the new highly sensitive troponin assays it has become clear that many patients have a troponin level above the 99th percentile when they have not suffered a myocardial infarction. We believe part of the problem with interpreting the the troponin values for patients is that the 99th percentile value which determines the ULN has been derived from population that is very different to the hospital population of patients. This study aims to demonstrate what the 99th percentile is for the population of people who use the hospital services who are traditionally older and have more comorbidities when compared to the population traditionally used to define the 99th percentile of a troponin assay.

An amendment was approved to follow-up patients' clinical outcomes at 1 year using NHS Digital data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older).
* Biochemistry blood sample already taken as part of routine clinical care.

Exclusion Criteria:

* Individuals aged less than 18 years old.
* No biochemistry blood sample taken as part of routine clinical care.
* Biochemistry samples requested by General Practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive patients (inpatients or outpatients) who have had a biochemistry sample requested by a hospital clinician as part of their routine clinical care. A total of 20,000 consecutive patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The 99th percentile for the hospital population. | 6 months
  Distribution and 99th centile for hsTnI BC assay in 20000 consecutive patients having a biochemistry blood test at a large teaching hospital

SECONDARY OUTCOMES:
The 99th percentile in different variables. | 6 months
  Distribution and 99th centile for hsTnI BC assay in:
  * Outpatients versus inpatients
  * Age by quintiles
  * Female vs male
  * ITU
  * General medicine inpatients: chest infection/exacerbation of COPD/PE/DVT/overdose etc
  * Emergency department, stratified by final diagnosis
  * General surgery
  * Major vascular surgery
  * Major abdominal surgery
  * Orthopaedic surgery… particularly fractured neck of femur and mortality outcome
  * Brain surgery
  * Rheumatoid outpatients according to level of disease activity
  * Autoimmune disease inpatients and outpatients
  * Inflammatory bowel disease inpatients & outpatients
  * COPD inpatients & outpatients
  * Diabetic outpatients and inpatients
  * Dermatology outpatients according to activity of disease (psoriasis/pemphigus etc)
The 99th percentile in different variables. | 12 months
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Nick Curzen, BM, PhD, Principal Investigator — Southampton NHS Trust
Locations (1):
- Southampton General Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariathas M, Allan R, Ramamoorthy S, Olechowski B, Hinton J, Azor M, Nicholas Z, Calver A, Corbett S, Mahmoudi M, Rawlins J, Simpson I, Wilkinson J, Kwok CS, Cook P, Mamas MA, Curzen N. True 99th centile of high sensitivity cardiac troponin for hospital patients: prospective, observational cohort study. BMJ. 2019 Mar 13;364:l729. doi: 10.1136/bmj.l729. PMID 30867154